CLINICAL TRIAL: NCT01138800
Title: Assessing Chronic Pain Conditions in Patients With and Without Interstitial Cystitis
Brief Title: Assessing Chronic Pain Conditions in Patients (Pts) With and Without (w&wo) Interstitial Cystitis
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-094
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Interstitial cystitis (IC) is a chronic disorder with significant symptoms of urinary urgency, frequency and pelvic pain. IC is more prevalent in women than men. Similar to other chronic pain syndromes such such as irritable bowel syndrome (IBS) and fibromyalgia, the cause of IC is not fully understood. Two subtypes of IC have been identified: classic IC (ulcerative IC) where visible ulcers exist in the bladder and non ulcerative IC, where bladder abnormalities are not apparent but significant bladder-related symptoms exist. We hypothesize that ulcerative IC is a disease of the bladder whereas non ulcerative IC is a more generalized and centrally-mediated chronic pain syndrome similar to IBS and fibromyalgia. To test this hypothesis, we will compare the presence of pain conditions/symptoms in ulcerative vs. non ulcerative IC women vs. community dwelling women (controls) without an IC diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age with IC identified by investigator (cases);
* Women over 18 years of age with IC (controls)

Exclusion Criteria:

* Male gender;
* subjects less than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 years of age with IC identified from the investigators practice (cases); women over 18 years of age without IC (controls)
Sampling Method: Probability Sample
Enrollment: 666 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital - Urology Research, Royal Oak, Michigan, United States